CLINICAL TRIAL: NCT02572960
Title: Physiologic Interactions Between the Adrenal- and the Parathyroid Glands
Acronym: AldOst
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-LSB
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2016-05

CONDITIONS: Osteoporosis; Vitamin D Deficiency; Cardiovascular Disease
MeSH Terms: conditions — Osteoporosis; Vitamin D Deficiency; Cardiovascular Diseases | interventions — Valsartan; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cholecalciferol (Placebo Comparator): Cholecalciferol 70 mcg/day for 12 weeks Placebo Valsartan daily for 2 weeks
  Interventions: Dietary Supplement: Cholecalciferol
- Valsartan (Active Comparator): Placebo cholecalciferol/day for 12 weeks Valsartan 80 mg/day for 2 weeks
  Interventions: Drug: Valsartan
- Placebo (Placebo Comparator): Placebo cholecalciferol/day for 12 weeks Placebo Valsartan daily for 2 weeks
  Interventions: Drug: Placebo Valsartan; Dietary Supplement: Placebo cholecalciferol
- Cholecalciferol and Valsartan (Active Comparator): Cholecalciferol 70 mcg/day for 12 weeks Valsartan 80 mg/day for 2 weeks
  Interventions: Drug: Valsartan; Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Drug: Valsartan — 2 weeks of Valsartan 80 mg per day
  Arms: Cholecalciferol and Valsartan; Valsartan
Drug: Placebo Valsartan — 2 weeks of Placebo Valsartan, one tablet per day. Placebo tablets are identical in regards to size and appearance to the experimental intervention tablet.
  Arms: Placebo
Dietary Supplement: Cholecalciferol — 12 weeks of daily cholecalciferol treatment, 70 microgram per day
  Other Names: Vitamin D3
  Arms: Cholecalciferol; Cholecalciferol and Valsartan
Dietary Supplement: Placebo cholecalciferol — 12 weeks of daily Placebo cholecalciferol treatment. Placebo tablets are identical in regards to size and appearance to the experimental intervention tablet.
  Other Names: Placebo D3
  Arms: Placebo

SUMMARY:
To investigate possible physiologic interactions between the adrenal- and the parathyroid glands in patients with secondary hyperparathyroidism.

DETAILED DESCRIPTION:
In primary hyperparathyroidism, chronic-elevated PTH levels seem to stimulate the renin-angiotensin-aldosterone system (RAAS) which may explain the increased risk of cardiovascular disease. In addition to increased PTH levels, vitamin D has been shown to inhibit the RAAS. However, a possible physiologic interaction needs further investigation.

The purpose of the study is to investigate changes in the RAAS in otherwise healthy postmenopausal women with secondary hyperparathyroidism due to vitamin D deficiency when p-PTH is normalized.

Furthermore, we will evaluate whether an angiotensin 2 receptor blocker can lower PTH in patients with secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Secondary hyperparathyroidism due to Vitamin D deficiency

Exclusion Criteria:

* Cardiovascular disease
* Renal failure
* Liver failure
* Treatment with antihypertensive medication or diuretics
* Treatment with lithium, NSAID or glucocorticoids
* Calcium supplement more than 500 mg per day or Vitamin D supplement more than 25 microgram per day
* Medical treatment for osteoporosis
* Systolic blood pressure below 120 mmHg
* Hypercalcaemia (more than 1,33mmol/L)
* Use of solarium or planned trip to countries, that might increase the endogenous vitamin D synthesis
* Allergic reaction to ACEi or ARBs.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Aldosterone, before and after 12 weeks of daily cholecalciferol treatment | Change from baseline p-aldosterone at 12 weeks

SECONDARY OUTCOMES:
Parathyroid hormone, before and after, daily ARB administrations | Change from baseline p-PTH at 2 weeks
Arterial stiffness | Change from baseline arterial stiffness at 12 weeks
  Spygmocor
24 hours arterial stiffness as measured by tonometry | Change from baseline arterial stiffness PWV at 12 weeks
  Arteriograph 24
24 hours blood pressure measured by tonometry | Change from baseline systolic pressure at 12 weeks
  Arteriograph 24
Balance as measured by stadiometer (Meitur Ltd) | Change from postural balance at 12 weeks
  Postural stability
Muscle strength as measured by isometric tests | Change from baseline isometric muscle strength at 12 weeks
  Effects on muscle strength (isometric tests of flexion and extension of thigh and hand), two function-tests (timed up-and go and timed stand-and-sit),
Bone density and geometry as measured by QCT scans | Change from baseline at 12 weeks
  Bone quality in spine and hip as assessed by high resolution quantitative computed tomography HRQCT-scans
Bone density and geometry as measured by HRpQCT scans | Change from baseline at 12 weeks
  Bone quality in ankle and forearm as assessed by high resolution peripheral quantitative computed tomography HRpQCT-scans
Bone density by DXA | Change from baseline at 12 weeks
  Bone density assessed by dual energy x-ray absorptiometry (DXA)
Electrocardiogram | Change from baseline at 2, 6 and 12 weeks
  Hearth rhythm, shortened QT interval, hypertrophy
Biomarkers of calcium- and bone metabolism | Change from baseline at 2, 6 and 12 weeks
  Effects of intervention on biochemical markers of calcium and bone metabolism, such as calcium, phosphate, parathyroid hormone, calcitriol, vitamin D-binding protein, bone-specific alkaline phosphatase, osteocalcin, and N-terminal propeptide of type 1 procollagen (P1NP). Also C-terminal telopeptide of type 1 collagen (CTX) and N-telopeptide of type 1 collagen (NTX) among others.
Quality of Life, SF36 | Change from baseline at 12 weeks
  SF36v2
Quality of Life, WHO-5 | Change from baseline at 12 weeks
  WHO-5 well being index
Physical activity | Change from baseline at 12 weeks
  Physical activity scale
Hyperparathyroid symptoms | Change from baseline at 12 weeks
  Pasieka's parathyroid symptoms score

CONTACTS AND LOCATIONS:
Overall Officials: Lars Rejnmark, Professor, Principal Investigator — Department of Endocrinology and Internal medicine
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bislev LS, Wamberg L, Rolighed L, Grove-Laugesen D, Rejnmark L. Effect of Daily Vitamin D3 Supplementation on Muscle Health: An Individual Participant Meta-analysis. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1317-1327. doi: 10.1210/clinem/dgac004. PMID 35018442
- [Derived] Bislev LS, Langagergaard Rodbro L, Rolighed L, Sikjaer T, Rejnmark L. Bone Microstructure in Response to Vitamin D3 Supplementation: A Randomized Placebo-Controlled Trial. Calcif Tissue Int. 2019 Feb;104(2):160-170. doi: 10.1007/s00223-018-0481-6. Epub 2018 Oct 6. PMID 30293198
- [Derived] Bislev LS, Langagergaard Rodbro L, Rolighed L, Sikjaer T, Rejnmark L. Effects of Vitamin D3 Supplementation on Muscle Strength, Mass, and Physical Performance in Women with Vitamin D Insufficiency: A Randomized Placebo-Controlled Trial. Calcif Tissue Int. 2018 Nov;103(5):483-493. doi: 10.1007/s00223-018-0443-z. Epub 2018 Jun 21. PMID 29931459